CLINICAL TRIAL: NCT05006287
Title: A Randomized Trial of the Safety of Non-vitamin K Oral Anticoagulants Compared to Warfarin Early After Cardiac Surgery: a Pilot Study
Brief Title: The Safety of Non-vitamin K Oral Anticoagulants Compared to Warfarin Early After Cardiac Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Jian Ye, MD, Cardiac Surgery, Clinical Professor, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StPaulH
Record Dates: First submitted 2021-05-29; First posted 2021-08-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation
Keywords: postoperative anticoagulation; warfarin; NOAC; cardiac surgery; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban; Dabigatran; edoxaban; Rivaroxaban; Warfarin

STUDY DESIGN:
Intervention Model Description: a multi-center, prospective, randomized, open-label, blinded-endpoint (PROBE) pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Vitamin K Oral Anticoagulant (NOAC) Group (Experimental): Anticoagulation with a NOAC (Apixaban, Dabigatran, Edoxaban, Rivaroxaban)
  Interventions: Drug: Non-vitamin K oral anticoagulants (NOACs)
- Warfarin Group (Active Comparator): Anticoagulation with warfarin to target INR 2.5
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Non-vitamin K oral anticoagulants (NOACs) — NOAC Group (Intervention):
  Patients randomized to the NOAC group will receive a NOAC dosed according to the Canadian monograph for the respective indication. Patients receiving a NOAC before cardiac surgery will resume the same NOAC as pre-operatively, whereas patients not previously receiving a NOAC will preferentially receive apixaban according to local practice. The NOAC will be started no earlier than post-operative day 5 and based on the standard protocol depending on whether the patient has a pre-existing indication for anticoagulation or new indication (e.g. post-operative atrial fibrillation).
  Patients at high risk of thrombosis and low risk of bleeding will receive a standardized bridging protocol as early as post-operative day 3 with unfractionated heparin infusion or low molecular weight heparin until the NOAC is initiated.
  Other Names: Apixaban, Dabigatran, Edoxaban, Rivaroxaban
  Arms: Non-Vitamin K Oral Anticoagulant (NOAC) Group
Drug: Warfarin — Warfarin Group (Comparator):
  Patients randomized to the warfarin group will receive warfarin titrated to achieve a target International Normalized Ratio (INR) of 2.5 (range 2.0 to 3.0). Warfarin will be started as early as post-operative day 1 and based on the standard protocol depending on whether the patient has a pre-existing indication for anticoagulation or new indication (e.g. post-operative atrial fibrillation).
  Patients at high risk of thrombosis and low risk of bleeding will receive a standardized bridging protocol as early as post-operative day 3 with unfractionated heparin infusion or low molecular weight heparin until INR is 2.0 or above.
  Arms: Warfarin Group

SUMMARY:
A small pilot study comparing different blood thinners (non-vitamin K oral anticoagulants [NOACs] and warfarin) will be conducted in people at risk for blood clots after open-heart surgery. This study will help us design a much bigger study to test the effectiveness and safety of different blood thinners in people after open-heart surgery. The study will test the following hypotheses: (1) Our standardized use of different blood thinners is feasible in patients early after cardiac surgery. (2) NOACs are safe to use early after cardiac surgery.

DETAILED DESCRIPTION:
Patients undergoing cardiac surgery (CVS) have various indications for anticoagulation, with the most common being pre-existing atrial fibrillation (AF) or post-operative atrial fibrillation (POAF). The incidence of POAF is up to 42% and both pre-existing AF and POAF have been associated with 62% higher odds of stroke and 44% higher odds of mortality. Even though non-vitamin K oral anticoagulants (NOACs) have superseded warfarin as the choice anticoagulant for non-valvular AF based on the results of landmark trials, these trials generally excluded patients with recent CVS. Although recommendations on anticoagulation for POAF are extrapolated from general AF guidelines, there is hesitancy to use NOACs early after cardiac surgery due to concerns regarding hemorrhagic cardiac tamponade and the fast anticoagulant onset of these agents with limited access to reversal agents. The investigators recently conducted a systematic review of 7 studies evaluating NOACs in the post-CVS setting, which identified insufficient evidence regarding the safety and efficacy of NOACs versus warfarin. Despite there being 3 planned randomized controlled trials (RCT) comparing NOACs to warfarin early following cardiac surgery, none indicated a standardized bridging protocol, which is a significant limitation, as anticoagulation trials lacking in standardized bridging may significantly influence incidences of bleeding and embolic events. The investigators propose a multi-centered pilot RCT of 100 patients comparing NOACs to warfarin initiated early after cardiac surgery (ie. within the index hospitalization) to determine the feasibility of conducting a large, definitive RCT. Patients with an indication for anticoagulation (most common being pre-existing AF or POAF), will be randomized to receive a NOAC (starting on post-operative day [POD] 5 or later) or warfarin (starting on POD 1 or at time of diagnosis of indication for anticoagulation) and supported by a standardized bridging protocol with unfractionated heparin infusion or low molecular weight heparin as early as POD 3 in patients with high-risk of thrombosis and low risk of bleeding. The co-primary feasibility outcomes are (1) >70% of eligible patients recruited into the study, and (2) >80% adherence to the anticoagulation protocol (defined as adherence to the bridging protocol and the initiation of the study drug on the right POD). The primary scientific outcome is a composite of death, stroke or systemic embolism, major bleeding, or pericardial effusion requiring intervention. Follow up will be conducted at 1 and 3 months and corroborated by re-admission data. The results of this pilot RCT will inform the design and feasibility of a large definitive RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years
2. Cardiac surgical procedures

   1. Coronary artery bypass grafting (on or off pump)
   2. Bioprosthetic aortic valve replacement
   3. Mitral valve repair
   4. Ascending aorta procedures
   5. Tricuspid valve repair
   6. Pulmonic valve procedures.
3. An indication for oral anticoagulation

   1. Pre-existing AF
   2. New post-operative atrial fibrillation
   3. Arterial embolism
   4. Venous thromboembolism.

Exclusion Criteria:

1. Cardiac surgical procedure

   1. Redo-sternotomy
   2. Bioprosthetic mitral valve replacement
   3. Mechanical valve replacement
   4. Transcatheter valve procedure
   5. Aortic arch procedures
   6. Pericardectomy
   7. Post-operative extracorporeal membrane oxygenation
   8. Heart transplant
   9. Ventricular assist devices
   10. Congenital heart procedures
2. Stroke within 4 weeks prior to surgery or postoperatively prior to initiation of study drug
3. Recent history of heparin-induced thrombocytopenia (less than 3 months)
4. High risk for bleeding (e.g. major bleed [intracranial hemorrhage, gastrointestinal bleed] within past 3 months, unexplained drop in hemoglobin pre-operatively)
5. Postoperative bleeding requiring return to operating room for exploration prior to randomization
6. Perioperative severe renal failure, defined as any eGFR <30 mL/min/1.73m2 or requirement of dialysis
7. Perioperative liver failure with alanine aminotransferase > 3x upper limit of normal
8. Pregnant or lactating women
9. Patient unable to consent
10. Contraindication to any study drug (including use of concomitant strong P-glycoprotein or cytochrome P450 enzyme inducers/inhibitors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Successful recruitment rate | At study completion (ie. 3 months)
  The percentage of eligible participants who can be successfully recruited in the study
Adherence rate to the anticoagulation protocol | At study completion (ie. 3 months)
  The percentage of participants who are adherent to the pre-specified anticoagulation protocol (ie. day of initiation of NOAC or warfarin, indication and dosing of bridging) during index hospital stay
Composite safety endpoint | 3 months
  The percentage of participants who experience all-cause mortality, major bleeding, stroke or systemic embolism, pericardial effusion requiring intervention

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No